CLINICAL TRIAL: NCT05945433
Title: Anovo™ Surgical System - Registry Study
Status: Recruiting | Type: Observational
Sponsor: Momentis Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: Momentis2023GYNRegistry
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: GYN Disorders
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients undergoing gynecological surgical procedure with the anovo Surgical System
  Interventions: Device: anovo™ Surgical System

INTERVENTIONS:
Device: anovo™ Surgical System — The anovo Surgical System is an endoscopic instrument control system that is intended to assist in the accurate control of the Instrument ARMS during single site, natural orifice laparoscopic-assisted transvaginal benign surgical procedures.

SUMMARY:
To collect Real-World Data (RWD) on the ongoing safety and effectiveness of the anovo Surgical system in transvaginal gynecological laparoscopic surgical procedures and to obtain information on the impact of the anovo Skills Development Pathway on user behavior and performance (where performance is measured by the learning curve of the surgeons and procedure outcomes).

DETAILED DESCRIPTION:
Specific Aims:

1. To collect RWD from surgeons with varying experience and expertise on their learning curve and time to achieve competency, and as such assess the success of the Skills Development Pathway.
2. Collect safety information and analyze the causality between type and frequency of adverse events to surgeons' experience.
3. Evaluate the effectiveness of the device while minimizing bias by enrolling "all comers", which will represent the general patient population.

ELIGIBILITY:
All patients receiving gynecological surgical procedure with the anovo Surgical System by their surgeon will be offered to participate in the registry.

Inclusion Criteria:

* patients must understand and sign the informed consent form, including data privacy authorization, indicating their consent to participate in the registry study.
* willing to complete post-operative questionnaire

Exclusion Criteria:

-none

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving gynecological surgical procedure with the anovo Surgical System by their surgeon will be offered to participate in the registry. To be eligible to participate in the registry, patients must understand and sign the informed consent form, including data privacy authorization, indicating their consent to participate in the registry study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Conversion rate to open or laparoscopic approach | Procedure
Rate of Unanticipated Adverse Device Effect | 8 Weeks Follow Up

SECONDARY OUTCOMES:
Surgery time (minutes) | Procedure

OTHER OUTCOMES:
Surgeon Learning Curve (surgery time against number of operations performed, considering frequency of cases and surgery difficulty) | Procedure
  To be reported as a continuous curve (plot per surgeon), and as the mean difference in surgery times between during learning curve and after learning curve stages (stages defined as before the surgeon achieves a steady state surgical time and after the surgeon achieves the steady state)
Surgeon Safety Curve (cumulative UADEs against number of operations performed) | Procedure
User Skills Development Survey | Procedure

CONTACTS AND LOCATIONS:
Locations (1):
- AdventHealth, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided